CLINICAL TRIAL: NCT05541692
Title: Efficacy of a Sleep Hygiene Toolkit for Patients in Acute Rehabilitation Unit
Brief Title: Efficacy of a Sleep Hygiene Toolkit for Patients in ARU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Joshua Kotler, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP-22-00115
Record Dates: First submitted 2022-09-02; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Sleep Disturbance; Sleep Disorder; Insomnia; Critical Illness Myopathy
Keywords: Occupational Therapy; Sleep; ARU; ADL; Rehab; sensory; cognitive behavior therapy; assistive devices; environmental disturbances
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficacy of a sleep hygiene toolkit in ARU (Other): Pre/post of intervention group (no control)
  Interventions: Behavioral: Sleep Hygiene Toolkit

INTERVENTIONS:
Behavioral: Sleep Hygiene Toolkit — The sleep hygiene toolkit includes multiple resources including assistive devices (ie. eye masks and ear plugs), sensory-based tools (ie. aromatherapy, music, meditation, and breathing techniques), cognitive behavioral therapy (CBT) activities (ie. addressing anxiety and worry), and education and training on sleep hygiene.

SUMMARY:
Sleep Hygiene Study Abstract:

INTRODUCTION Sleep is integral to the health of a person and can have multifaceted contributions to a person including their physical, cognitive, and psychosocial well-being. However, within a recent survey evaluating the sleep perception of patients within an acute rehabilitation unit (ARU), there was a high prevalence of reported sleep disturbances and poor sleep hygiene compared to at home (Davis et al., 2021). In addition, patients within an ARU generally have an extended length of stay-which could mean many nights of poor sleep hygiene. Given the importance of sleep in facilitating a person's health and recovery versus the challenges the hospital environment poses on patient's sleep hygiene, this study aims to examine the efficacy of a sleep hygiene toolkit provided to the patients admitted to ARU. The sleep hygiene toolkit includes multiple non-pharmaceutical resources addressing sensory stimulation and psychological and emotional needs.

OBJECTIVE This study aims to evaluate the perception of sleep quality experienced by ARU patients utilizing the sleep hygiene toolkit. This study hypothesizes that with the use of a sleep hygiene toolkit, patients will report a positive impact on their sleep quality during their hospital stay.

METHODOLOGY This is a within-subjects study design. All eligible participants will be given the sleep hygiene intervention administered for a period of five days. The sleep hygiene toolkit includes multiple resources including assistive devices (ie. eye masks and ear plugs), sensory-based tools (ie. aromatherapy, music, meditation, and breathing techniques), cognitive behavioral therapy (CBT) activities (ie. addressing anxiety and worry), and education and training on sleep hygiene. The visual analog scales on the Richards-Campbell Sleep Questionnaire will be used to assess patient's overall sleep perception pre- and post-intervention.

CONCLUSION Given this prevalent area of need for patients admitted to ARU, occupational therapists (OT) can offer an additional way to address it. According to the Occupational Therapy Practice Framework (2020), OTs are well-equipped to provide comprehensive treatment to promote a person's sleep preparation and sleep participation. The results will determine the efficacy of a sleep hygiene toolkit for ARU patients in addressing their sleep needs-an important component in a patient's health and recovery during their hospital stay.

SIGNIFICANCE OF TOPIC This study aims to highlight the barriers to successful participation in the occupation of sleep and rest for patients admitted to an acute rehabilitation unit (ARU). The creation of this sleep hygiene toolkit is to address a person's sleep preparation and sleep participation. Although sleep quality and its impact are a topic well studied, there is limited study on occupational therapy led interventions aimed to benefit the patient's sleep quality in an ARU setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have the ability and willingness to give informed consent
* ability to communicate verbally and understand the questionnaires
* ability to use all components of the intervention
* are expected to stay in ARU for more than five days.

Exclusion Criteria:

* Patients with severe cognitive, communication, or behavioral deficits
* received a score of 7 or less out of 15 on the Brief Interview for Mental Status (BIMS) upon admission
* unable to use all components of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire | 5 days
  Visual analog scale aimed to assess patient's overall sleep perception. Scale parameters are from 0-100 with the higher number correlating to better sleep perception. This questionnaire was used pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Medical Center of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Publication of data analysis related to intervention study findings